CLINICAL TRIAL: NCT01115088
Title: Effects of Stevia on Satiety and Eating Attitudes in Healthy, Overweight and Obese Adults: A Pilot Study
Brief Title: Effects of Stevia on Satiety and Eating Attitudes in Healthy, Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, William Cefalu, MD, Executive Director, Pennington Biomedical Research Center
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: PBRC 25030
Record Dates: First submitted 2010-04-29; First posted 2010-05-04 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Aspartame; Sucrose; stevioside

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aspartame (Experimental): Food or beverages containing Aspartame in comparison to Stevia or Sucrose
  Interventions: Dietary Supplement: Aspartame
- Sucrose (Experimental): Food or beverages containing Sucrose in comparison to Aspartame or Stevia
  Interventions: Dietary Supplement: Sucrose
- Stevia (Experimental): Food or beverages containing Stevia in comparison to Aspartame or Sucrose
  Interventions: Dietary Supplement: Stevia

INTERVENTIONS:
Dietary Supplement: Aspartame — The morning breakfast after a 12-h fast and consumed a standard 469 kcal breakfast consisting of cereal, milk, toast with butter, and orange juice. Tea and crackers with cream cheese sweetened with stevia Whole Foods 365 Brand, aspartame equal sweetener, or sucrose participants consumed this preload 20 min before their test lunch and dinner meals. The Test lunch meal consisted of sandwiches, potato chips, and cookies, and the test dinner meal was a self-selected buffet-type meal (I.e., Macronutrient Self-Selection Paradigm) Geiselman et al,. 1998)
  Other Names: equal sweetener
  Arms: Aspartame
Dietary Supplement: Sucrose — The morning breakfast after a 12-h fast and consumed a standard 469 kcal breakfast consisting of cereal, milk, toast with butter, and orange juice. Tea and crackers with cream cheese sweetened with stevia Whole Foods 365 Brand, aspartame equal sweetener, or sucrose participants consumed this preload 20 min before their test lunch and dinner meals. The Test lunch meal consisted of sandwiches, potato chips, and cookies, and the test dinner meal was a self-selected buffet-type meal (I.e., Macronutrient Self-Selection Paradigm) Geiselman et al,. 1998)
  Arms: Sucrose
Dietary Supplement: Stevia — The morning breakfast after a 12-h fast and consumed a standard 469 kcal breakfast consisting of cereal, milk, toast with butter, and orange juice. Tea and crackers with cream cheese sweetened with stevia Whole Foods 365 Brand, aspartame equal sweetener, or sucrose participants consumed this preload 20 min before their test lunch and dinner meals. The Test lunch meal consisted of sandwiches, potato chips, and cookies, and the test dinner meal was a self-selected buffet-type meal (I.e., Macronutrient Self-Selection Paradigm) Geiselman et al,. 1998)
  Arms: Stevia

SUMMARY:
The purpose of this study is to test the effects that three different types of sweeteners have on food intake, hunger and satiety levels, as well as insulin and glucose measures. The study of whether food or beverages containing Stevia influence food intake to a greater extent than food or beverages sweetened with Aspartame or Sucrose. Also, examining whether taste preference and taste sensitivity influence food intake.

DETAILED DESCRIPTION:
Expected time in this study will be approximately 24 hours spread over the course of one initial screening visit and three test days during which you complete food tests at the Pennington Center.

Screening visit (Duration is 3 hours)

* You will initially be asked to fill out psychological questionnaires to assess your eating habits, food cravings, and preference for foods (i.e., tea and crackers with cream cheese) that will be provided to you in this study.
* You will also be asked to complete two taste tests during this visit. The first taste test will be sodium chloride (table salt) followed by PROP (an extremely low dose of hyperthyroid medication) sodium chloride (table salt).
* You will be required to provide a blood sample (19 mL or 1.3 tablespoons) to check glucose and insulin levels.
* If you are selected to be a participant for this study, you will receive a brief medical evaluation during which you will be weighed, your height will be measured, and your pulse and blood pressure will be taken. You will be interviewed about your medical history and potential obstacles for completing the study. If you are female, a brief interview will be conducted to determine your menstrual cycle phase. Total length of time will be approximately three hours for the screening visit.

First Food Test Day (Duration is 7- 9 hours. You'll arrive after having fasted for 12 hrs.) For females, all test meal days will be scheduled during their luteal phase. • Breakfast: During your first food test day, you will be asked to come to the Pennington Center at any time between the hours of 7:00 A.M. - 8:30 A.M. and consume a standard breakfast of Cheerios, milk, orange juice, toast, butter, and jelly. You will then be free to leave but will be asked to return 3.5 hours later. When your return, you will be sent to our inpatient unit for a blood draw, which will test your level of insulin and glucose (total of 25 mL or 1.67 tablespoons). You will then be asked to rate your appetite on a computer using a visual analog scale (VAS). After completing these VAS ratings, you will be provided with an appetizer of 5 ounces of cold tea and 6 crackers with cream cheese. Both the tea and the cream cheese will be sweetened with one of the following sweeteners: Aspartame, Sucrose, or Stevia. After consuming this appetizer, you will be asked to complete another set of VAS ratings, which again ask you about your appetite, as well as the sweetness of the appetizer. Test times will be constant for all visits. Approximately twenty minutes after consuming this appetizer, your insulin and glucose levels will again be tested and you will complete another set of VAS ratings before your lunch meal. You will be required to consume breakfast at the same time for all three visits. For example, if you come at 7:00 A.M. on your first test day, you will be required to come in at 7:00 A.M. on your next two test days.

• Lunch: After completing VAS ratings before lunch, you will be provided with a lunch consisting of sandwiches, chips, and cookies. Your lunch meal will be served approximately 4 hours after your breakfast meal. Your eating behavior may be monitored by weight of the food consumed and/or by video camera/tape. You may eat as much or as little of the lunch as you wish.

• After Lunch: After you finish your lunch meal, you will be asked to complete post meal VAS ratings. Your insulin and glucose will be measured on the three occasions after lunch: 30 minutes after lunch, one hour after lunch, and two hours after lunch for a total of 5 blood draws (total of 25 mL or 1.67 tablespoons). You will also be asked to complete VAS ratings 30 minutes after lunch, and every hour for the next four hours. You will spend the afternoon at the Pennington center to ensure that blood draws and VAS ratings occur at the appropriate time intervals. During the afternoon you will be free to read, do paperwork brought from home or work, or watch movies that will be provided to you by the Center.

• Dinner:

Four hours after the test lunch, you will be provided with another appetizer of 5 ounces of cold tea and crackers with cream cheese. Both the tea and the cream cheese will be sweetened with one of the following sweeteners: Stevia, sucrose, or Aspartame. You will complete VAS ratings before and after this appetizer, as well as before and after your dinner meal (4.5 hours after lunch), during which you will be instructed to eat as much or as little of any of the items presented as you want. Your eating behavior may be monitored by weight of the food consumed and/or by video camera/tape. After you complete VAS questions after the evening meal, you will have fulfilled the requirements of the first food test day. However, you will be asked not to consume any food or caloric beverages for three hours following your dinner meal. You will be asked to report any adverse events from this day at this visit.

Second Food Test Day (Duration is 7-9 hours. You'll arrive after having fasted for 12 hrs.) • On your second food test day, you will complete the same procedures and meal tests as you did during the first food test day. However, the type of sweetener used in your tea and crackers with cream cheese will differ from the type of sweetener you received on your first food test day. You will be asked to report any adverse events from this day, as well as previous visits, at this visit.

Third Food Test Day (Duration is 7-9 hours. You'll arrive after having fasted for 12 hrs.)

• On your third food test day, you will complete the same procedures and meal tests as you did during your two previous food test days. However, the type of sweetener used in your tea and crackers with cream cheese will differ from the type of sweetener you received on previous visits. You will also be asked to report any adverse events from this day, as well as previous visits, at this visit. We will also follow up by phone regarding adverse events following your third visit. Table 1 presents a schedule of the procedures that will take place at each of the study visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and have a body mass index > 30 kg/m2 and < 39.9 kg/m2, or have a body mass index > 20 kg/m2 and < 24.9 kg/m2
* If BMI is between 30 and 39.9, waist circumference must be > 36 for women and > 40 for men.
* Age 18 to 45 years
* Nonsmokers
* Willing to consume meat products
* Women on monophasic oral contraceptives or who have physiologically controlled cycles

Exclusion Criteria:

* A history of diabetes, cardiovascular disease, or other chronic illnesses
* Presence of an eating disorder including Anorexia and/or Bulimia Nervosa
* Other health problems that might interfere with your ability to participate in the study
* Taking medications, other than monophasic birth control or monophasic (same dose every day) hormone replacement therapy and allergy medication
* Taking allergy medication for a period of time less than 6 months
* Dislike of or allergy to foods/sweeteners (Sucrose, Stevia, or Aspartame) used in test meals
* Smokers
* High scores on the Dietary Restraint, Disinhibition, and Perceived Hunger scales of the Three Factor Eating Questionnaire
* Use of oral contraceptives other than monophasic (same dose every day) contraceptives

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Effects of stevia, aspartame, and sucrose on food intake, satiety, and postprandial glucose and insulin levels. | 24 hours
  Test whether preloads of tea and crackers with cream cheese sweetened with Stevia lover postprandial insulin levels compared to preloads of tea and crackers with cream cheese sweetened with Sucrose or Aspartame by measuring blood insulin and glucose levels immediately prior to the lunch preload,immediately before lunch test meal, and at thirty minutes, one hour, and two hours after the lunch test meal.

SECONDARY OUTCOMES:
Hedonic ratings (appearance, aroma, flavor, texture and palatability)with Stevia sweetener compared to Sucrose or Aspartame | 24 hours
  Test whether preloads of tea and crackers with cream cheese sweetened with Stevia have different hedonic ratings compared to preloads of tea and crackers with cream cheese sweetened with Sucrose or Aspartame by examining hunger and satiety ratings after the preload.
Satiating effects by examining food consumption | 24 Hours
  Test whether preloads of tea and crackers with cream cheese sweetened with stevia have different satiating effects compared to preloads of tea and crackers with cream cheese sweetened with Sucrose or Aspartame by examining food consumption 20 minutes and after lunch and dinner preloads, as well as total food consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Anton, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States